CLINICAL TRIAL: NCT05567965
Title: Live Better at Home (Catalonia): a Randomized Clinical Trial
Brief Title: Live Better at Home in Catalonia
Acronym: VMCat
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Vic - Central University of Catalonia (Other)
Collaborators: Spanish Society of Geriatrics and Gerontology (Unknown)
Responsible Party: Principal Investigator, Eduard Minobes, Doctor, University of Vic - Central University of Catalonia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VMCCat1.0
Record Dates: First submitted 2022-09-27; First posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-09

CONDITIONS: Geriatrics; Home Care Services
Keywords: Older people; Home care; Functional capacity; Dependence

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensified home care intervention + Training (Experimental): Users will receive an intensification in their home care intervention for dependence, receiving an intervention of a minimum of 1 hour per day and a maximum of 3.5 hours, to support their activities of daily living. The intensification will be personalised according to the specific needs of the user that the professionals consider necessary to attend. The weekly distribution of the intervention will be flexible in terms of timetables, as agreed between professional and informal caregivers. In addition, each informal caregiver will receive multimodal online training with the aim of providing knowledge, skills and attitudes that empower them to face the challenge of caring, guaranteeing quality care, preventing situations that may negatively affect both the person and the family dynamics and enabling an optimal evolution in caregiving.
  Interventions: Other: Home care intervention
- Conventional home care intervention (Active Comparator): Participants will continue with their conventional home care intervention for dependence, comprising activities that are mainly carried out at the users' home and are oriented towards supporting their activities of daily living. This intervention is of personalised attention and its average intensity is about 20 minutes per day.
  Interventions: Other: Home care intervention

INTERVENTIONS:
Other: Home care intervention — The duration of the intervention, both for the control group and the intervention group, will be 18 months or until the user's admission to the nursing home.

SUMMARY:
The intensity of the home care interventions for dependent older people offered in Spain, and specifically in Catalonia, may not be sufficient to help keep older people at home and delay institutionalisation in a nursing home, but an intensification of the intervention could improve the health and psychosocial state of dependent people and their informal caregivers and facilitate their permanence at home.

DETAILED DESCRIPTION:
According to recent surveys, more than 80% of older people prefer to live at home, so the current model of care should aim to prolong the autonomy of older people so that they remain as long as possible at home and delay their entry into nursing homes.

The hypothesis of the study is that an intensification of the home care intervention in users with degree II or III of dependency will delay or avoid their institutionalisation in nursing homes.

The main aim of the study is to evaluate the effect of an intensification in home care interventions on users with grade II or III dependency in order to delay or avoid their institutionalisation in a geriatric residence.

Secondary aims are to analyse the effect of an intensification of home care interventions in users with degree II or III of dependency on their health and psychosocial state.To analyse the effect of an intensification of home care intervention together with training for informal caregivers on the health status and overburden of informal caregivers of users with degree II or III of dependency.

To test the impact on the use of resources of an intensification of home care interventions in users with degree II or III of dependency.

A randomised clinical trial with two parallel arms and blinded assessment will be conducted. The duration of follow-up will be 18 months. It will be carried out at the community level in homes in eight municipalities in the province of Barcelona, Catalonia (Spain).

ELIGIBILITY:
Inclusion Criteria:

* Older people (men and women aged 65 and over).
* Living in the community.
* Categorized with a degree II or III of dependency.
* Users of the public home care without requesting admission to an institution in Catalonia.
* With a main informal caregiver in charge.
* The acceptance to participate in the study of the user and the informal caregiver.

Exclusion Criteria:

* Users with privately paid professional carers.
* Users in palliative care (short life expectancy).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change in time from baseline until application for nursing home admission | Every month up to 18 months. Assessed from the baseline in the study until the application for entry in nursing home, assessed up to 18 months.
  To the user. Assessed by asking.

SECONDARY OUTCOMES:
Functional capacity | Every 3 months up to 18 months.
  To the user. Assessed by the Barthel Index. The scoring range is 0 (total dependency)-100 (slight dependency)
Frailty | Every 3 months up to 18 months.
  To the user. Assessed by the Frail-VIG index. The scoring range is 0 (no frailty)- 25 (advanced frailty).
Risk of sarcopenia | Every 3 months up to 18 months.
  To the user. Assessed by the strength, assistance with walking, rising from a chair, climbing stairs, and falls (SARC-F) questionnaire. The scoring range is 0 - 10 (more than 4 points means risk of sarcopenia).
Risk of falls | Every 3 months up to 18 months.
  To the user. Assessed by the Downton Scale. The scoring range is 0 - 14 (more than 3 points means risk of falls).
Cognitive status | Every 3 months up to 18 months.
  To the user. Assessed by the Reisberg Global Deterioration Scale. The scoring range is 1 (no dementia)- 7 (late-stage dementia).
Social network | Every 3 months up to 18 months.
  To the user. Assessed by the Lubben Social Network Scale. The scoring range is 0 (less social engagement)- 30 (more social engagement).
Chronic patient experience | Every 3 months up to 18 months.
  To the user. Assessed by the Chronic Patient Experince Evaluation Instrument (IEXPAC). The scoring range is 0 (worst experience)- 110 (best experience).
Quality of life related with health | Every 1 month up to 18 months.
  To the user. Assessed by the EUROQOL-5D-3L. The scoring range is 0 (worst quality of life)- 100 (best quality of life).

OTHER OUTCOMES:
Physical activity grade | Every 3 months up to 18 months.
  To the informal caregiver. Assessed by the International Physical Activity Questionnaire-Short Form (IPAQ). The classification ranges from low level of physical activity to high level of physical activity.
Caregiver overburden | Every 3 months up to 18 months.
  To the informal caregiver. Assessed by the Zarit Burden Scale. The scoring range is 5 (no overburden)- 35 (more overburden).
Experience of the informal caregiver with people with chronic disease | Every 3 months up to 18 months.
  To the informal caregiver. Assessed by the Chronic Patient Experince Evaluation Instrument for caregivers(IEXPAC caregivers). The scoring range is 0 (worst experience)- 120 (best experience).

CONTACTS AND LOCATIONS:
Overall Officials: Jose Augusto Garcia Navarro, Principal Investigator — Spanish Society of Geriatrics and Gerontology

IPD SHARING:
Plan to Share IPD: Yes
All collected data will result in some publications
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication
Access Criteria: Access criteria will be made on demand

REFERENCES:
- [Derived] Minobes-Molina E, Pamies-Tejedor S, Roncal-Belzunce V, Escalada San Adrian G, Atares Rodriguez L, Garcia-Navarro JA. Multimodal home care intervention for dependent older people "Live better at home": Protocol of a randomized clinical trial. Rev Esp Geriatr Gerontol. 2023 Jul-Aug;58(4):101383. doi: 10.1016/j.regg.2023.101383. Epub 2023 Jul 13. PMID 37453249